CLINICAL TRIAL: NCT04825860
Title: A Randomized, Double-blind, Parallel-group, Placebo Controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of SEP 363856 in Acutely Psychotic Patients With Schizophrenia, Followed by an Open-label Extension Phase
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic People With Schizophrenia, Followed by an Open-label Extension Phase
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to company business strategy
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA801201; jRCT2071210003 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEP-363856 50 mg/day (Experimental): Subjects randomized to the SEP-363856 50 mg/day group will receive the assigned dose of SEP-363856 50 mg/day throughout the double-blind phase.
  Interventions: Drug: SEP-363856 50 mg
- SEP-363856 75 mg/day (Experimental): Subjects randomized to the SEP-363856 75 mg/day group will receive SEP-363856 50 mg/day on Day 1 through Day 3 and then the assigned dose of SEP-363856 75 mg/day thereafter.
  Interventions: Drug: SEP-363856 75 mg
- Placebo (Placebo Comparator): Subjects randomized to the placebo group will receive placebo throughout the double-blind phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 50 mg — Subjects will take one tablet of study drug per day at approximately the same time each evening at bedtime. Study drug may be taken orally with or without food.
  Arms: SEP-363856 50 mg/day
Drug: SEP-363856 75 mg — Subjects will take one tablet of study drug per day at approximately the same time each evening at bedtime. Study drug may be taken orally with or without food.
  Arms: SEP-363856 75 mg/day
Drug: Placebo — Subjects will take one tablet of study drug per day at approximately the same time each evening at bedtime. Study drug may be taken orally with or without food.
  Arms: Placebo

SUMMARY:
A clinical study to investigate the effect of 2 doses of an investigational drug in acutely psychotic adult patients with schizophrenia. The study will consist of a double-blind phase followed by an open-label extension phase.

DETAILED DESCRIPTION:
A Phase 2/3 Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Patients with Schizophrenia, Followed by an Open-label Extension Phase.

The double-blind phase is to evaluate the efficacy and safety of 2 doses of SEP-363856 (50 and 75 mg/day) versus placebo over 6 weeks in acutely psychotic patients with schizophrenia. This phase is projected to randomize approximately 480 subjects to 3 treatments (SEP-363856 50 mg/day, SEP-363856 75 mg/day, placebo) in a 1:1:1 ratio. The completers of the double-blind phase will be able to enroll into the 12-week open-label phase during which the long term safety and effectiveness of-SEP 363856 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Must be fully informed of and understand the objectives, procedures, and possible benefits and risks of the study, and give written informed consent prior to performing any study related activities. If the subject is considered a minor according to local regulations at the time of collection of the informed consent, written consent will be obtained from a legally acceptable representative (guardian) in addition to that obtained from the subject.
2. Male or female between 18 to 65 years of age (inclusive) at the time of consent.
3. Must meet DSM 5 criteria for schizophrenia as established by clinical interview at Screening
4. Must have a CGI S score ≥ 4 (moderately ill) at Screening and Baseline.
5. Must have a PANSS total score ≥ 80 and a PANSS item score ≥ 4 (moderate) on 2 or more of the following PANSS items: delusions (P1), conceptual disorganization (P2), hallucinations (P3), and unusual thought content (G9) at Screening and Baseline.
6. Must have an acute exacerbation of psychotic symptoms (no longer than 2 months prior to providing informed consent for this study). The acute exacerbation should include:

   a. Marked deterioration of functioning in one or more areas, such as occupational, social, or personal care or hygiene.
7. In the opinion of the Investigator, subjects must be generally healthy based on Screening medical history, physical examination (PE), vital signs, ECG, and clinical laboratory values (hematology, chemistry, and urinalysis).

Exclusion Criteria:

1. Have a DSM 5 diagnosis or presence of symptoms consistent with a DSM 5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months, or lifetime history of significant substance abuse that, in the opinion of the Investigator, may have had a significant and potentially permanent impact on the brain or other body systems, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder, and posttraumatic stress disorder. Symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms have not been a focus of primary treatment
2. At significant risk of harming self, others, or objects based on Investigator's judgment.
3. Have any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study.
4. Female subjects who are pregnant or lactating.
5. Have any clinically significant abnormal laboratory value(s) at Screening (hematology, chemistry, and urinalysis) as determined by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Positive and negative syndrome scale (PANSS) total score at Week 6 | Week 6
  PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impressions - Severity (CGI-S) score at Week 6 | Week 6
  The CGI-S is a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.

CONTACTS AND LOCATIONS:
Locations (54):
- China (8):
  - Beijing Anding Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second People's Hospital of Hunan Province/ Brain Hospital of Hunan Province, Changsha, Hu'nan
  - Shandong Daizhuang Hospital, Jining, Shandong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - The Mental Health Center of Xi'an, Xian, Shanxi
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
- Japan (38):
  - Hotei Hospital, Kōnan, Aichi-ken
  - Okehazama Hospital Fujita Kokoro Care Center, Toyoake, Aichi-ken
  - Medical corporation Seijinkai Seinan Hospital, Hachinohe, Aomori
  - Kohnodai Hp., National Center for Global Health and Medicine, Ichikawa, Chiba
  - Shiranui Hospital, Omuta, Fukuoka
  - Juzenkai Oorin Hospital, Ōnojō, Fukuoka
  - Takeda General Hospital, Aizu-Wakamatsu, Fukushima
  - Mihara Hospital, Mihara, Hiroshima
  - Fujimidai Hospital, Hiratsuka, Kanagawa
  - Okinawa Tokushukai Hino Hospital, Yokohama, Kanagawa
  - Yatsushiro Kosei Hospital, Yatsushiro, Kumamoto
  - Miyakonojo Shinsei Hospital, Miyakonojō, Miyazaki
  - Shonan Hospital, Matsumoto, Nagano
  - Mental Support Soyokaze Hospital, Ueda, Nagano
  - NHO Ryukyu Hospital, Kunigami, Okinawa
  - Social welfare corporation Tenshinkai Kosaka hospital, Higashiosaka, Osaka
  - Kansai Medical University Medical Center, Moriguchi, Osaka
  - Nishiurakai Keihan Hospital, Moriguchi, Osaka
  - Neyagawa Sanatorium, Neyagawa, Osaka
  - Asakayama Hospital, Sakai, Osaka
  - Osaka Institute of Clinical Psychiatry Shin-abuyama Hospital, Takatsuki, Osaka
  - NHO Hizen Psychiatric Center, Kanzaki, Saga-ken
  - Rainbow & Sea Hospital, Karatsu, Saga-ken
  - Nishi Kumagaya Hospital, Kumagaya, Saitama
  - Shiga university of medical science hospital, Ōtsu, Shiga
  - Negishi Hospital, Fuchū, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Narimasu Kosei Hospital, tabashi City, Tokyo
  - National Hospital Organization Hokuriku National Hospital, Nanto, Toyama
  - Azusakai Kawada Hospital, Takaoka, Toyama
  - Sanyokai Sanyo Hospital, Sakata, Yamagata
  - Akino Hospital, Tendō, Yamagata
  - Akita City Hospital, Akita
  - Inokuchi Noma Hospital, Fukuoka
  - Kuramitsu Hospital, Fukuoka
  - Minkodo Aburayama Hospital, Fukuoka
  - Satokai Yuge Hospital, Kumamoto
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
- Philippines (5):
  - Mariveles Mental Wellness and General Hospital, Mariveles, Bataan
  - St. Paul's Hospital of Iloilo, Inc., Iloilo City, Iloilo
  - Makati Medical Center, Makati City, National Capital Region
  - National Center for Mental Health, Mandaluyong, National Capital Region
  - Southern Philippines Medical Center, Davao City
- Taiwan (3):
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No